CLINICAL TRIAL: NCT01973179
Title: Observational Study to Re-irradiation for Recurrent Head and Neck Cancer
Brief Title: Re-irradiation of Recurrent Head and Neck Cancer
Acronym: ReKo
Status: Active, not recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Mechthild Krause, Prof. Dr. med., Technische Universität Dresden
Other Study IDs: STR-ReKo-2013
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2024-01

CONDITIONS: Head-and-neck Carcinoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiation therapy: Radiotherapy with protons in patients with head and neck carcinoma
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy with protons

SUMMARY:
The goal of this observational study is to evaluate the toxicity and local tumor control of proton therapy for patients with head and neck cancer in a previously irradiated field.

Standard of care for recurrent or secondary malignancies in a previously irradiated field is surgery. For inoperable patients or residual tumor after surgery, standard of care would be palliative chemotherapy. For a small subset of patients (good performance status, small radiation fields) re-irradiation can be performed. In this study the established concept of re-irradiation with photons will be transferred to proton radiotherapy. Proton therapy has the advantage of a steeper dose gradient to normal tissues, thus-theoretical advantages for lower toxicity.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary: Evaluation of late toxicity of re-irradiation with protons, for patients with head and neck cancer in a previously (> 50 Gy) irradiated field.

Secondary: Evaluation of the efficacy (local control) and acute toxicity (after 24 Months) of re-irradiation with protons up to a dose of 60 Gy, for patients with head and neck cancer in a previously (> 50 Gy) irradiated field.

OUTLINE This is a single center observational study. In-house standard of care for patients (good performance status and with small tumors) with head and neck cancer in a previously (> 50 Gy) irradiated field is to irradiate the tumor with a hyperfractionated schedule and concurrent cisplatin up to a dose of 66 Gy. Dose limiting for this schedule is the incidence of acute and late toxicity induced by radiation. The purpose of the study is the evaluation of the safety of a treatment schedule based on the use of protons.

Proton beam treatments will be delivered in 2 Gy fractions, 5 days per week, to a total dose of 60-66 Gy equivalent.

Study visits are performed:

During proton therapy once per week. Follow-up visits are scheduled every 3 months for the first 24 months after proton therapy.

Primary endpoint is late toxicity 24 months after proton treatment.

ELIGIBILITY:
Inclusion Criteria:

* tumor is located in a previously irradiated area with at least 50 Gy or there is an overlap of radiation fields with resulting total doses greater than 90 Gy to expect
* tumor size and localization allow high dose re-irradiation (individual decision)
* exclusion of distant metastases
* Time interval between pre-irradiation and re- irradiation at least 1 year for local recurrence; at least 6 months for secondary tumor disease
* age ≥ 18 years
* previous radiotherapy treatment plans available
* pre-treatment imaging (pre re-irradiation) available
* good general condition (ECOG 0-1)
* dental treatment performed, if necessary
* in case of surgery before re-irradiation: resection status is R-1 or R-2
* clinical suspicion of residual tumor by very scarce surgical margins (<1 mm)
* pathological secured extracapsular extension (ECE)
* indications by an interdisciplinary tumor board
* patient able to understand the intention and procedures of the trial, written informed consent

Exclusion Criteria:

* no description of the R- status after resection of the tumour
* pregnancy
* no written informed consent
* distant metastases
* interval between first and second irradiation < 6 months at secondary tumor or <1 year when local recurrence of previously irradiated tumor
* simultaneous participation in another intervention study , if further treatment must be carried out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a recurrent or secondary head and neck carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
late toxicity | 24 months after therapy
  measured from the first day of treatment

SECONDARY OUTCOMES:
acute toxicity | 3 months after treatment
  measured from the first day of treatment
local recurrence free survival | 24 months after therapy
  measured from the first day of treatment
overall survival | 24 months after therapy
  measured from the first day of treatment
quality of life | 24 months after therapy
  measured from the first day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mechthild Krause, Prof., Study Chair — Dresden University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology; and DKTK partner site Dresden
Locations (1):
- Dresden University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology; and DKTK partner site Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No